CLINICAL TRIAL: NCT04275531
Title: Evaluation of Possible Neurotoxicity of Anesthesia Guided by Olfactory Changes in Middle-aged Patients
Brief Title: Neurotoxicity of Anesthesia in Middle Aged Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Raafat Elghamry, principal investigator, Tanta University
Other Study IDs: neurotoxicity of anesthesia
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia; Adverse Effect
MeSH Terms: interventions — Anesthetics; Sevoflurane; Isoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- regional anesthesia: surgical procedures which will be performed under intrathecal anesthesia without sedation
  Interventions: Drug: Anesthesia Agent
- sevoflurane: surgical procedures which will be performed under general anesthesia and sevoflurane will be used for maintenance of anesthesia
  Interventions: Drug: Anesthesia Agent
- isoflurane: surgical procedures which will be performed under general anesthesia and isoflurane will be used for maintenance of anesthesia
  Interventions: Drug: Anesthesia Agent
- propofol: surgical procedures which will be performed under general anesthesia and propofol infusion will be used for maintenance of anesthesia
  Interventions: Drug: Anesthesia Agent

INTERVENTIONS:
Drug: Anesthesia Agent — various anesthetic agents used in both general and regional anesthesia
  Other Names: Sevoflurane; Isoflurane; Propofol infusion

SUMMARY:
for the last 20 years, the increasing reports from non-human studies have raised suspicion that general anesthetics may cause neurotoxic changes in the developing brain that lead to adverse neurodevelopmental outcomes later in life.there are several case reports of reversible smell and taste dysfunction following exposure to general anesthesia suggesting a possible relationship between anesthetic agents and olfactory dysfunction.

this study is to assess the possible neurotoxicity of sevoflurane,isoflurane,and propofol based anesthesia guided by olfactory changes

DETAILED DESCRIPTION:
the primary inhibitory neurotransmitter GABA is found in neuronal synapses involving olfactory bulb. So, the involvement of common GABA pathway implies a possible interaction of general anesthetics with olfactory function.

olfactory identification is an associative memory which is found to be facilitated by action of melatonin. involvement of GABA receptor in the transfer of light information from suprachiasmatic nuclei to pineal gland suggests possible interaction of melatonin and anesthetic agents.

the aim of the study is to evaluate the possible neurotoxicity of sevoflurane,isoflurane,and propofol based anesthesia guided by olfactory changes

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-50 years
* both sex
* American society of Anesthesiologists' physical status I and II
* elective surgery of duration 90-120 minutes

Exclusion Criteria:

* patients's refusal
* recent airway infection
* allergic rhinitis
* nasal polyps
* history of alcoholism
* smoking
* pregnancy
* menstruating female
* mental retardation
* psychiatric illness
* neurosurgical or oto-rhino-laryngeal surgery
* history of olfactory deficits or cognitive impairment
* CNS disease e.g. epilepsy
* history of first degree relative with alzheimer's disease,dementia, or cognitive dysfunction
* those who are unable to answer the tests themselves

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: middle aged patients, of both sex, undergoing elective surgical procedures other than major surgeries, of duration 90-120 minutes, and of American Society of Anesthesiologists' physical status I and II will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
olfactory threshold | olfactory threshold will be measured at 12 hours preoperative then at 6, 24 and 48 hours postoperative
  we will use (10 dilutions) of 4% n-butyl alcohol. The odorant and a blank will be presented to the participant. The test will be progressed from weaker-to-stronger concentrations of odorant. Two bottles will be presented to each participant, an odorant bottle and an identical bottle filled with distilled water. The participant will sniff each one for 9 seconds and then will chose which one smelled stronger. If the participant is incorrect at one concentration, the next higher concentration will be presented. When the correct choice is made, the same concentration of odorant will be presented to the participant until four consecutive correct responses are given.

SECONDARY OUTCOMES:
olfactory identification | Smell identification will be measured at 12 hours preoperative then at 6, 24 and 48 hours postoperative
  We will use UPSIT test.
cognitive dysfunction | Cognitive dysfunction will be evaluated at 12 hours preoperative then at 6, 24 and 48 hours postoperative
  cognitive dysfunction will be evaluated by mini-mental state examination
serum melatonin concentrations | serum melatonin will be measured at 12 hours preoperative then at 6, 24 and 48 hours postoperative
  Melatonin levels will be measured in plasma by the enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Elghamry, MD, Principal Investigator — Tanta University, Faculty of Medicine
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
statistics of demographic data,type of surgeries, olfactory dysfunction tests,mini-mental state examination, and serum melatonin
Supporting Information: SAP
Time Frame: Individual patient data will be shared after finishing and publication of the study and it will be available for 6 months.
Access Criteria: the individual patient data will be available for scientific research only up on email request. request will be sent to email of principal investigator (drmonagh19802000@gmail.com)